CLINICAL TRIAL: NCT01323491
Title: Nicht-interventionelle Studie (NIS) Zur Strukturierten Raucherentwöhnung Nach Dem Konzept "EINFACH ERFOLGREICH RAUCHFREI" unterstützt Durch NICROETTE®-Produkte
Brief Title: "EASY EFFECTIVE SMOKELESS" With NICORETTE®
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson GmbH (Industry)
Collaborators: Anfomed GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: EER Nicorette - 01
Record Dates: First submitted 2011-03-21; First posted 2011-03-25 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Stereotyped Behavior; Tobacco Smoking Behavior
Keywords: smoking cessation; nicotine replacement therapy; routine smokers
MeSH Terms: conditions — Stereotyped Behavior; Smoking; Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- routine smokers: would-be non-smokers, no actual nicotine replacement therapy
  Interventions: Drug: Nicotine replacement therapy

INTERVENTIONS:
Drug: Nicotine replacement therapy — Nicorette® TX tape 10mg, 15mg, 25mg Nicorette® microtab 2mg Nicorette® inhaler 10mg Nicorette® chewing gum 2 mg, 4mg freshfruit, freshmint, mint, whitemint

SUMMARY:
The actually most accepted method of effective smoking cessation is based on structured consultation and medical care in combination with supportive medical treatment. A group of experts developed the concept "EINFACH ERFOLGREICH RAUCHFREI" ("EASY EFFECTIVE SMOKELESS") for general practitioners providing a structured compendium for negotiation.

Physicians who have implemented this concept will conduct this non-interventional study. The implementation of the scheme will be investigated under general practice conditions and the applicability of the concept has to be assessed by the physicians.

In addition further knowledge of smoking cessation in would-be non-smokers which decided to quit, supported by medical treatment with NICORETTE®-products, will be documented for a large patient collective under real practice conditions.

To answer all above mentioned questions for a sufficient number of patients a multicenter, prospective non-interventional study design was used for this trial as only this instrument detects characteristics of the physicians' treatment without any further input or other influences.

ELIGIBILITY:
Inclusion Criteria:

* Routine smokers
* Nicotine replacement therapy with Nicorette® according to physicians treatment decision

Exclusion Criteria:

* Pregnancy
* Contraindication according to Summary of Product Characteristics (SPC)
* Other nicotine replacement therapy during the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: general practitioners
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2011-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Further knowledge of smoking cessation in would-be non-smokers | Baseline (about 2 weeks before date of smoking cessation), Follow-up (about 3, 14 and 28 days after date of smoking cessation), Final examination (about 3 months after date of smoking cessation)

CONTACTS AND LOCATIONS:
Locations (1):
- Johnson & Johnson GmbH, Neuss, Germany